CLINICAL TRIAL: NCT02927704
Title: Gingival Crevicular Fluid Levels Of Monocyte Chemoattractant Protein-1 in Patients With Aggressive Periodontitis
Brief Title: Gingival Crevicular Fluid Levels Of Monocyte Chemoattractant Protein-1
Acronym: MCP-1
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Collaborators: Selcuk University (Other)
Responsible Party: Principal Investigator, Sadiye Gunpinar, Abant Izzet Baysal University Faculty of Dentistry periodontology department, Abant Izzet Baysal University
Other Study IDs: 2011/016; 11102024 (Other Grant/Funding Number: Selcuk University Scientific Foundation); konya2013 (Other: last day of the study)
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Aggressive Periodontitis
Keywords: Aggressive Periodontitis; monocyte chemoattractant protein-1; gingival crevicular fluid; enzyme-linked immunosorbent assay
MeSH Terms: conditions — Aggressive Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- case (Aggressive periodontitis): Single intervention has been performed for each subject. Gingival crevicular fluid sample was obtained in conjunction with clinical measurements in this intervention.
  Interventions: Other: Gingival crevicular fluid (GCF) sample
- control (Periodontally healthy subjects): Single intervention has been performed for each subject. Gingival crevicular fluid sample was obtained in conjunction with clinical measurements in this intervention.
  Interventions: Other: Gingival crevicular fluid (GCF) sample

INTERVENTIONS:
Other: Gingival crevicular fluid (GCF) sample — Single intervention has been performed for each subject. GCF samples were collected from four multi rooted teeth (premolar/molar) one of in each quadrant including two maxilla and two mandibula by single examiner in conjunction with clinical measurements in this intervention.

SUMMARY:
The aim of this study is to estimate GCF MCP-1 levels of healthy and Aggressive periodontitis (AgP) subjects and to compare MCP-1 levels between Localized AgP (LAgP) and Generalized AgP (GAgP) to establish its predictive value/role for distinguishing LAgP and GAgP development.

DETAILED DESCRIPTION:
Patients with aggressive periodontitis (AgP) are diagnosed as rapid and severe periodontal destruction commonly in younger systemically healthy individuals (Armitage, 1999). Although periopathogenic bacteria are essential for initiation, this alone does not be responsible for the manifestation and severity of the clinical status/phenotype (Offenbacher et al., 2008), suggesting an imbalance between host and bacterial load (Kinane et al., 2007). Response to bacterial biofilm is determined by the host immune system (Mahanonda and Pichyangkul, 2007, Amano, 2010) in which genetic and enviromental factors modify and may get individuals more susceptible or resistant to the periodontal diseases (Kulkarni and Kinane, 2014).

The role of whether an impaired or a hyperinflammatory host response is responsible for the progression of aggressive periodontitis has been a topic of discussion. Regarding to this topic Shaddox et al. (2016) studied the whole blood specimens collected from LAgP subjects and stimulated with plaque sample generated from healthy or diseased sites. And as a result, LAgP subjects displayed hyperinflammatory response regardless of contents of bacterial stimulus. In an another research hyperinflammatory responders LAgP subjects presented the lowest reductions in clinical parameters, on the contrary low responders showed the highest reductions after treatment (Allin et al., 2016). Similarly Garrison and Nichols (1989) reported that hyper-inflammatory monocyte phenotype can be deterministic in periodontal destruction. In the view of the aforementioned findings, the aim of this study is to estimate GCF MCP-1 levels of healthy and AgP subjects and to compare MCP-1 levels between LAgP and GAgP to establish its predictive value/role for distinguishing LAgP and GAgP development.

A total of 160 subjects including, 80 AgP and 80 age and gender matched periodontally healthy (H) controls were recruited in this cross-sectional study. Clinical periodontal measurements including plaque index (PI), gingival index (GI), proping depth (PD) and clinical attachment loss (CAL) were performed. GCF samples were collected from 160 patients including 50 LAgP, 30 GAgP and 80 H. Volume of GCF samples were measured by an electronic device (Periotron 8000, OroFlow Inc.) and GCF MCP-1 was measured by an enzyme-linked immunosorbent assay "ELISA".

ELIGIBILITY:
Inclusion Criteria:

* Periodontally Healthy control group (n: 80) had < 3mm PD, < 2 GI and no signs of interproximal attachment loss and a history of periodontal disease.
* The AgP group included individuals diagnosed with localized AgP (LAgP) or generalized AgP (GAgP) who were otherwise healthy. Periodontal attachment loss ≥4 mm accompanied by interproximal bone loss without gingival recession not involving more than two permanent teeth, other than the first molars and incisors were diagnosed with LAgP (n: 50); patients with involvement of at least three teeth, other than the first molars and incisors with an attachment loss ≥4 mm accompanied by interproximal bone loss without gingival recession were diagnosed with GAgP (n: 30).

Exclusion Criteria:

* Patients who have any systemic diseases or conditions that could effect the periodontium
* hepatitis and/or immunodeficiency virus infection
* a history of periodontal treatment and antibiotic therapy within the 6 months
* < 16 teeth in their mouth
* Subjects who had smoked and were ongoing orthodontic treatment were excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This cross-sectional case control study was carried out at Selcuk University, Faculty of Dentistry, Department of Periodontology. Aggressive periodontitis patients referred as case were diagnosed by single examiner.The control group included periodontally healthy volunteers from staff and other subjects referring to the School of Dentistry.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2011-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Determination of GCF MCP-1 levels in patients with AgP | 1 year

SECONDARY OUTCOMES:
Measurement of clinical periodontal parameters in patients with AgP and compare between LAgP and GAgP | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sadiye Gunpinar, Asst. Prof., Principal Investigator — Abant Izzet Baysal University, Faculty of Dentistry, Periodontology Department; Nilgun O Alptekin, Prof., Principal Investigator — Baskent University, Faculty of Dentistry, Periodontology Department; Niyazi Dundar, Dr., Principal Investigator — Selcuk University, Faculty of Dentistry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armitage GC. Periodontal diagnoses and classification of periodontal diseases. Periodontol 2000. 2004;34:9-21. doi: 10.1046/j.0906-6713.2002.003421.x. No abstract available. PMID 14717852
- [Background] Lee E, Yang YH, Ho YP, Ho KY, Tsai CC. Potential role of vascular endothelial growth factor, interleukin-8 and monocyte chemoattractant protein-1 in periodontal diseases. Kaohsiung J Med Sci. 2003 Aug;19(8):406-15. doi: 10.1016/S1607-551X(09)70484-X. PMID 12962428
- [Background] Kurtis B, Tuter G, Serdar M, Akdemir P, Uygur C, Firatli E, Bal B. Gingival crevicular fluid levels of monocyte chemoattractant protein-1 and tumor necrosis factor-alpha in patients with chronic and aggressive periodontitis. J Periodontol. 2005 Nov;76(11):1849-55. doi: 10.1902/jop.2005.76.11.1849. PMID 16274303
- [Background] Gupta M, Chaturvedi R, Jain A. Role of monocyte chemoattractant protein-1 (MCP-1) as an immune-diagnostic biomarker in the pathogenesis of chronic periodontal disease. Cytokine. 2013 Mar;61(3):892-7. doi: 10.1016/j.cyto.2012.12.012. Epub 2013 Jan 30. PMID 23375122
- [Background] Emingil G, Atilla G, Huseyinov A. Gingival crevicular fluid monocyte chemoattractant protein-1 and RANTES levels in patients with generalized aggressive periodontitis. J Clin Periodontol. 2004 Oct;31(10):829-34. doi: 10.1111/j.1600-051X.2004.00584.x. PMID 15367184
- [Background] Thunell DH, Tymkiw KD, Johnson GK, Joly S, Burnell KK, Cavanaugh JE, Brogden KA, Guthmiller JM. A multiplex immunoassay demonstrates reductions in gingival crevicular fluid cytokines following initial periodontal therapy. J Periodontal Res. 2010 Feb;45(1):148-52. doi: 10.1111/j.1600-0765.2009.01204.x. Epub 2009 Jul 8. PMID 19602112
- [Background] Tymkiw KD, Thunell DH, Johnson GK, Joly S, Burnell KK, Cavanaugh JE, Brogden KA, Guthmiller JM. Influence of smoking on gingival crevicular fluid cytokines in severe chronic periodontitis. J Clin Periodontol. 2011 Mar;38(3):219-28. doi: 10.1111/j.1600-051X.2010.01684.x. Epub 2010 Dec 29. PMID 21198766